CLINICAL TRIAL: NCT05753540
Title: Pilot Study on the Effects of MLS (Multiwave Locked System) LASER Therapy in Patients With Chronic Nonspecific Neck Pain: Randomized Controlled Trial Versus Placebo
Brief Title: The Effects of MLS LASER Therapy in Patients With Chronic Nonspecific Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Lisa Berti, Assistant, Istituto Ortopedico Rizzoli
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MLS LASER-neck
Record Dates: First submitted 2022-06-28; First posted 2023-03-03 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-05

CONDITIONS: Chronic Non-specific Neck Pain
MeSH Terms: interventions — Laser Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser therapy (Experimental): Multiwave locked system laser therapy
  Interventions: Other: Laser therapy
- Sham laser therapy (Placebo Comparator): Sham laser therapy
  Interventions: Other: Sham laser therapy

INTERVENTIONS:
Other: Laser therapy — Multiwave locked system laser therapy
  Arms: Laser therapy
Other: Sham laser therapy — Sham laser therapy
  Arms: Sham laser therapy

SUMMARY:
Non-specific cronic low back pain is very common condition affecting 30-50% of adults. It is featured by neck muscles contractures which lead to pain and reduction of cervical spine mobility. High intensity laser therapy has been shown to be an effective treatment to improve symothoms in patient with non-specific neck pain.

The aim of this study is to assess the effects of a multi-wave locked system laser therapy in patient with non-specif neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Chronic low back pain (> 3 months)
* Body mass index < 30
* Preserved cognitive ability to fully understand and observe indications received by medical personnel
* Ability to understand and give an informed consent

Exclusion Criteria:

* Spine surgery
* Spinal hernia
* spondylolisthesis
* Spinal infections
* Severe spine deformities
* Neural diseases
* Upper limbs radiculopathy
* Cervical rib
* Rotator cuff or other shoulder diseases
* Rheumatic diseases
* Diabetes
* Psychiatric diseases
* Vascular diseases
* Cancer
* Infectious diseases
* Skin abrasion
* Pregnancy or breastfeeding
* Recent injuries
* Known sensibility to Laser therapy
* Epilepsy
* Anticoagulant therapy
* Pacemaker
* hemorrhagic diathesis
* Photosensitizing drugs
* Known Photosensibility
* Neck Tattoos

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Change in Neck pain | Change from baseline neck pain at 3 and 7 weeks
  Eleven point (0-10) visual analogue scale

SECONDARY OUTCOMES:
Change in Disability | Change from baseline disability at 3 and 7 weeks
  Neck disability index questionnaire

OTHER OUTCOMES:
Change in Neck mobility | Change from baseline neck mobility at 3 and 7 weeks
  Degree of head rigth/left flexion, forward/backward flexion and rigth/left rotation, together with the velocity of the movements measured with an accelerometer

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Italy